CLINICAL TRIAL: NCT02292342
Title: An Acute, Double-blind, Randomised, Placebo-controlled, Crossover Intervention Trial Investigating the Dose-dependent Vascular Effects of Pure (-)-Epicatechin (≤1 mg/kg BW) in Healthy Men.
Brief Title: An Investigation of the Dose-dependent Vascualr Effects of (-)-Epicatechin in Healthy Men
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor Jeremy P.E. Spencer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EpicatechinStudy
Record Dates: First submitted 2014-10-23; First posted 2014-11-17 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Vasodilation
Keywords: Flow mediated dilatation
MeSH Terms: conditions — Aneurysm | interventions — Water; Catechin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.1 mg/ kg BW pure (-)-epicatechin (Active Comparator): 0.1 mg/ kg BW pure (-)-epicatechin (according to volunteer) dissolved in 3 ml/kg BW of water.
  Interventions: Dietary Supplement: Water; Dietary Supplement: Epicatechin 0.1 mg/kg; Dietary Supplement: Epicatechin 0.5 mg/kg; Dietary Supplement: Epicatechin 1.0 mg/kg
- 0.5 mg/ kg BW pure (-)-epicatechin (Active Comparator): 0.5 mg/ kg BW pure (-)-epicatechin (according to volunteer) dissolved in 3 ml/kg BW of water.
  Interventions: Dietary Supplement: Water; Dietary Supplement: Epicatechin 0.1 mg/kg; Dietary Supplement: Epicatechin 0.5 mg/kg; Dietary Supplement: Epicatechin 1.0 mg/kg
- 1.0 mg/ kg BW pure (-)-epicatechin (Active Comparator): 1.0 mg/ kg BW pure (-)-epicatechin (according to volunteer) dissolved in 3 ml/kg BW of water.
  Interventions: Dietary Supplement: Water; Dietary Supplement: Epicatechin 0.1 mg/kg; Dietary Supplement: Epicatechin 0.5 mg/kg; Dietary Supplement: Epicatechin 1.0 mg/kg
- 0.0 mg/ kg BW pure (-)-epicatechin (Placebo Comparator): Water only (3 ml/kg BW)
  Interventions: Dietary Supplement: Water; Dietary Supplement: Epicatechin 0.1 mg/kg; Dietary Supplement: Epicatechin 0.5 mg/kg; Dietary Supplement: Epicatechin 1.0 mg/kg

INTERVENTIONS:
Dietary Supplement: Water — Control
Dietary Supplement: Epicatechin 0.1 mg/kg — EC 0.1 mg/kg
Dietary Supplement: Epicatechin 0.5 mg/kg — EC 0.5
Dietary Supplement: Epicatechin 1.0 mg/kg — EC 1.0

SUMMARY:
Aim: To investigate the dose-dependent vascular effect (primarily using FMD) of 3 low-level doses of pure (-)-epicatechin ≤ 1 mg/kg BW (0.1, 0.5 & 1.0 mg/kg BW) in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 20-27.5 kg/m2
* Normal blood pressure at screening (< 150/90)
* Non-smoker
* Non-vegetarian
* 'Normal - low' chocolate consumer (<2 potions per week)
* 'Normal - low' coffee/ tea drinker (<3 cups per day)
* Regular exercise routine
* Signed consent form

Exclusion Criteria:

* Haemoglobin (anaemia marker) < 125 g/l
* Gamma GT (liver enzymes) > 80 IU/l
* Cholesterol > 6.5 mmol/l
* Suffered a myocardial infarction or stroke in the last 12 months
* Suffers from any cardiovascular or metabolic disorders (e.g. diabetes or any other endocrine or liver diseases)
* Suffers from any blood-clotting disorder, and/or takes supporting medication
* Any dietary restrictions or on a weight reducing diet
* On any lipid-modifying or blood pressure lowering medication
* Consuming any specific vitamin/ herbal supplements or fish oils

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | baseline to 2h

SECONDARY OUTCOMES:
Laser Doppler Imaging with Iontophoresis | baseline to 2h
Plasma (-)-epicatechin metabolites | baseline to 24h
Plasma nitrate/nitrite | baseline to 2h

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No